CLINICAL TRIAL: NCT04987944
Title: A Phase 1b, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate Safety and Efficacy of Oral Zavegepant in Subjects With Mild Allergic Asthma
Brief Title: Safety and Efficacy Active Drug vs. Placebo in Subjects With Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision to discontinue the study based on adjusted clinical development plan. This decision is not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BHV3500-204; C5301005 (Other: Alias Study Number)
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-02

CONDITIONS: Asthma
Keywords: Allergy; Asthma
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BHV3500 (Experimental): Zavegepant 150 mg BID
  Interventions: Drug: Zavegepant
- Placebo (Placebo Comparator): Matching placebo 150 mg BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zavegepant — 150 mg BID
  Other Names: BHV3500
  Arms: BHV3500
Drug: Placebo — Placebo matching active drug
  Arms: Placebo

SUMMARY:
This study is a double-blind, parallel-group, randomized study of active drug vs placebo in asthma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Asthma

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - The Lung Centre- Vancouver General Hospital, Vancouver, British Columbia
  - The Lung Centre-Vancouver General Hospital, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - McMaster Universtiy, Hamilton, Ontario
  - Institut universitaire en cardiologie et pneumologie de Quebec-Universite Laval-(IUCPQ-UL), Québec, Quebec
  - University of Saskatchewan/Royal University Hospital, Saskatoon, Saskatchewan
  - Institut universitaire en cardiologie et pneumologie de Quebec-Universite Laval-(IUCPQ-UL), Québec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3500-204

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 participants signed the informed consent form and were enrolled, of which 30 were screen failures and 15 participants were randomized into the study.
Groups:
- Zavegepant: Participants with mild allergic asthma, with a history of episodic wheeze and shortness of breath were administered 150 milligrams (mg) of zavegepant twice daily (BID) for 28 days. Participants were followed for up to 10 days post last dose of study treatment.
- Placebo: Participants with mild allergic asthma, with a history of episodic wheeze and shortness of breath were administered placebo BID for 28 days. Participants were followed for up to 10 days post last dose of study treatment.
Period: Overall Study
Arm/Group | Zavegepant | Placebo
Started | 7 | 8
Completed | 7 | 6
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zavegepant | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (14.40) | 29.3 (11.06) | 32.7 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percentage Decrease From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Any Time Between 3 and 7 Hours Post-Allergen Challenge
Description: Allergen inhalation challenge was performed on Day 27 and FEV1 was measured using spirometry prior to the challenge and between 3 to 7 hours post allergen challenge to assess late asthmatic response (LAR). FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. The maximum percentage decrease was the difference between the baseline (pre-allergen challenge) FEV1 on Day 27 and lowest FEV1 between hours 3 and 7 on Day 27 divided by the baseline value from Day 27. Analysis was performed using analysis of covariance (ANCOVA) model with treatment as main effect and baseline FEV1 as covariate.
Time Frame: Baseline (pre-allergen challenge on Day 27) and anytime between 3 and 7 hours post-challenge on Day 27
Population: Modified Intent-to-Treat (mITT) analysis set included participants who received at least 1 dose of study therapy and provided at least 1 non-missing post-baseline LAR assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 7 | 6
Percent change | 19.7 [9.9 to 29.5] | 29.5 [18.8 to 40.1]
Statistical Analysis 1: Comparison: Zavegepant vs Placebo; Test type: Other; Least square mean difference = -9.8, 95% CI 2-sided [-24.5 to 5.0]

2. Secondary Outcome: Maximum Percentage Decrease From Baseline in FEV1 at Any Time Between 0 and 2 Hours Post-Allergen Challenge
Description: Allergen inhalation challenge was performed on Day 27 and FEV1 was measured using spirometry prior to the challenge and between 0 to 2 hours post allergen challenge to assess early asthmatic response (EAR). FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. The maximum percentage decrease was the difference between the baseline (pre-allergen challenge) FEV1 on Day 27 and lowest FEV1 between hours 0 and 2 on Day 27 divided by the baseline value from Day 27. Analysis was performed using ANCOVA model with treatment as main effect and baseline FEV1 as covariate.
Time Frame: Baseline (pre-allergen challenge on Day 27) and anytime between 0 and 2 hours post-challenge on Day 27
Population: mITT analysis set included participants who received at least 1 dose of study therapy and provided at least 1 non-missing post-baseline LAR assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 7 | 6
Percent change | 30.5 [20.1 to 40.8] | 34.4 [23.2 to 45.5]
Statistical Analysis 1: Comparison: Zavegepant vs Placebo; Test type: Other; Least square mean difference = -3.9, 95% CI 2-sided [-19.4 to 11.5]

3. Secondary Outcome: Change in Methacholine PC20 From Pre-Allergen Challenge to Post-Allergen Challenge
Description: Airway hyperresponsiveness was assessed using methacholine provocation concentration causing a 20% decline in FEV1 (PC20). Change in PC20 from pre-allergen to post-allergen = PC20 in post-allergen challenge minus PC20 in pre-allergen challenge. Shift in PC20 was calculated as post-allergen challenge minus pre-allergen challenge (Day 28 minus Day 26), and baseline shift in PC20 was calculated as post-allergen challenge minus pre-allergen challenge (Day -13 minus Day-15). Analysis was performed using ANCOVA model with treatment as main effect and baseline shift as covariate.
Time Frame: From Day -15 to Day 28
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Milligrams per milliliter
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 7 | 6
Milligrams per milliliter | 0.165 [-0.192 to 0.521] | -0.259 [-0.671 to 0.154]
Statistical Analysis 1: Comparison: Zavegepant vs Placebo; Test type: Other; Least square mean difference = 0.423, 95% CI 2-sided [-0.125 to 0.972]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered an investigational (medicinal) product and that did not necessarily have a causal relationship with this treatment. An SAE was defined as any adverse event that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; life-threatening; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect or other important medical events. TEAEs were events with onset dates on or after the start of the study drug.
Time Frame: From start of treatment on Day 1 up to Day 41
Population: The safety analysis set included all randomized participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 7 | 8
Participants
  TEAEs | 3 | 4
  TESAEs | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities on Treatment
Description: The following laboratory parameters were assessed: hematology (eosinophils, hemoglobin, leukocytes, lymphocytes, neutrophils and platelets), chemistry (Albumin, alanine aminotransferase [ALT], alkaline phosphatase [ALP], aspartate aminotransferase [AST], bicarbonate, bilirubin, calcium, cholesterol, creatine kinase, creatinine, glucose, low-density lipoproteins [LDL], lactate dehydrogenase, potassium, sodium, triglycerides) and urinalysis (urine glucose and urine protein). Clinically significant laboratory test abnormalities were Grade 3 (severe) to Grade 4 (potentially life-threatening) laboratory test results graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 except for glucose, LDL cholesterol, uric acid and urinalysis which were graded using Division of Aids (DAIDS) Version 2.1 where, Grade 3=severe and Grade 4=potentially life-threatening. Number of participants with clinically significant abnormalities in any laboratory parameter is presented.
Time Frame: From start of treatment on Day 1 to Day 28
Population: The safety analysis set included all randomized participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: On treatment: From start of study treatment on Day 1 up to Day 28 and Follow up: From Day 29 to Day 41
Groups:
- Zavegepant (On Treatment): Participants with mild allergic asthma, with a history of episodic wheeze and shortness of breath were administered 150 milligrams (mg) of zavegepant twice daily (BID) for 28 days.
- Placebo (On Treatment): Participants with mild allergic asthma, with a history of episodic wheeze and shortness of breath were administered placebo BID for 28 days.
- Zavegepant (Follow-up): Participants who received zavegepant during treatment phase were followed for up to 10 days post last dose of study treatment.
- Placebo (Follow-up): Participants who received placebo during treatment phase were followed for up to 10 days post last dose of study treatment.
Arm/Group | Zavegepant (On Treatment) | Placebo (On Treatment) | Zavegepant (Follow-up) | Placebo (Follow-up)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 3/7 | 4/8 | 0/7 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant (On Treatment) (N=7) | Placebo (On Treatment) (N=8) | Zavegepant (Follow-up) (N=7) | Placebo (Follow-up) (N=8)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04987944/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04987944/SAP_001.pdf